CLINICAL TRIAL: NCT00967395
Title: Effect of Healing on Rheumatoid Arthritis: a Three-arm Double-blind, Randomized, Controlled Trial
Brief Title: Effect of Healing on Rheumatoid Arthritis
Acronym: RAhealing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henning Bliddal (Other)
Collaborators: The IMK Foundation (Unknown); The Danish Rheumatism Association (Other); Oak Foundation (Other)
Responsible Party: Sponsor-Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: (KF) 01-123/04; (KF) 01-123/04
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healing (Experimental): patients receive healing while blindfolded and with hearing protector. The healer is behind a screen and not allowed to speak with the subject.
  Interventions: Other: Healing
- Sham healing (Sham Comparator): Same design of room as with the healing, while in this case a student is behind the screen
  Interventions: Other: Sham healing
- Control (No Intervention): Business as usual in the third arm

INTERVENTIONS:
Other: Healing — Healing in our study is given be a healer "no-touch", who just has to be present in the room.
  Other Names: "active healing"
  Arms: Healing
Other: Sham healing — Sham Healing in our study is given be a student "no-touch", who just has to be present in the room.
  Other Names: "placebo healing"
  Arms: Sham healing

SUMMARY:
The hypothesis is that healing may influence the patient's general status by altering psychological as well as other body functions of importance for the rheumatoid arthritis. This is tested in a three group design with a control group and two groups receiving healing with or without a healer present. The study is randomized and double blind.

DETAILED DESCRIPTION:
The central claim of healers is that this process facilitates self-healing in the patient. Spiritual healing includes several categories, including 'therapeutic touch' and 'intercessory prayer', and the healing may be attributed to God, spirits, universal forces or energies, biological healing energies residing in the healer, or self-healing powers or energies thought to reside latent in the healed organism. The highly controversial hypothesized effects of distant or spiritual healing contradict our traditional sense of reality and are in conflict with what is generally viewed as being in correspondence with modern science.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis in a stable medication the past 3 months written informed consent

Exclusion Criteria:

* Not able to arrange own transport, language problems

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
DAS28 | 8 weeks follow-up

SECONDARY OUTCOMES:
Colour Doppler fraction | 8 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bente Danneskiold-Samsøe, Professor, Study Director — Frederiksberg University Hospital